CLINICAL TRIAL: NCT06306352
Title: The Effect of Vibrotactile Feedback on Exoskeleton Use in People With Motor Complete Spinal Cord Injury
Brief Title: Vibrotactile Feedback in Exoskeletons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Collaborators: ABLE Human Motion S.L. (Industry); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1070; NL82999.091.22 (Other: CCMO)
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injuries
Keywords: Exoskeletons; Sensory substitution; Vibrotactile feedback; Motor control; Motor learning
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibrotactile feedback (Experimental): Participants will receive vibrotactile feedback in the ABLE Exoskeleton.
  Interventions: Other: Vibrotactile feedback

INTERVENTIONS:
Other: Vibrotactile feedback — The ABLE exoskeleton is accompanied by a vibrotactile feedback belt which users wear around their chest to receive real-time feedback during the double support phase. This feedback can assist them in their weight shift during the double support phase.

SUMMARY:
This study aims to investigate the impact of providing discrete vibrotactile feedback related to weight shift and step initiation on exoskeleton use in individuals with motor-complete SCI.

DETAILED DESCRIPTION:
Rationale: People with motor-complete spinal cord injury (SCI) lack motor function below the lesion level and are, thus, wheelchair-dependent. In recent years, wearable exoskeletons have emerged as potential mobility devices for this population. Although exoskeletons generate the basic motions for ambulation, postural stability must be maintained by the user. People with motor-complete SCI miss essential somatosensory perception, which affects their ability to maintain postural stability. Hence, walking in an exoskeleton is demanding, and crutches are necessary.

When sensory information of a specific system is lost, the lack of sensory information can be substituted by providing feedback to another sensory system. As sensory feedback has been shown to improve postural control in people missing essential sensory information, such sensory substitution may also be effectively incorporated in people with complete SCI using an exoskeleton.

Objective: The study aims to investigate the effect of vibrotactile feedback on exoskeleton use in people with motor-complete SCI.

Study design: The proposed study is an experimental study. The study protocol includes six sessions of 90 minutes spread over three weeks. Sessions one to five are dedicated to training to assess the effect of vibrotactile feedback on exoskeleton motor learning. Session six is dedicated to evaluation to assess the effect of vibrotactile feedback on exoskeleton motor control.

ELIGIBILITY:
Inclusion Criteria:

* SCI classification American Spinal Injury Association Impairment Scale (AIS) A or B
* Minimally six months post-injury
* Prior experience with the ReWalk Exoskeleton, able to walk independently

Exclusion Criteria:

* Pre-existing somatosensory problems before the SCI
* Visual or auditory issues that are not resolved with glasses or a hearing device
* Insufficient mastery of the Dutch language
* Contraindications related to the ABLE Exoskeleton

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Walking distance covered | Up to 3 weeks
  Walking distance covered during a 50-second walking trial.

SECONDARY OUTCOMES:
Reach path ratio | Up to 3 weeks
  The reach path ratio of the Center of Mass (COM) trajectory in the double support phase.
Reach time | Up to 3 weeks
  The reach time represents the time spent in the double support phase.
User experience questionnaire | After 3 weeks
  A customized questionnaire to assess the specific user experience of the vibrotactile feedback system, considering key aspects related to exoskeleton motor learning and motor control. The questionnaire comprises five visual analog questions employing a scale ranging from strongly disagree to strongly agree
Dutch version of the Quebec User Evaluation of Satisfaction with Assistive Technology (D-QUEST) - only including the eight items related to user satisfaction with the assistive device | After 3 weeks
  The D-QUEST evaluates a patient's satisfaction with various assistive technologies.

OTHER OUTCOMES:
Dutch System Usability Scale (D-SUS) | After 3 weeks
  The SUS is a questionnaire-based method to assess the usability of a system or product through a series of standardized questions.

CONTACTS AND LOCATIONS:
Overall Officials: Noël Keijsers, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No